CLINICAL TRIAL: NCT00283283
Title: Clinical Study to Compare the Immune Response of Half Dose Trivalent Inactivated Influenza Vaccine (TIV) to Full Dose
Brief Title: Comparison of Full-dose Flu Vaccine to Half-dose Flu Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency); United States Army Medical Materiel Development Activity (U.S. Federal Agency); Centers for Disease Control and Prevention (U.S. Federal Agency); Uniformed Services University of the Health Sciences (U.S. Federal Agency); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); U.S. Air Force Office of the Surgeon General (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A-13205
Record Dates: First submitted 2006-01-24; First posted 2006-01-27 (Estimated); Results first posted 2020-06-19 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (8):
- Male, Age 18 -49, Full Dose (Experimental): 0.5ml, 15µg Fluzone® (Aventis Pasteur inactivated influenza vaccine) hemagglutinin antigen per strain
  Interventions: Biological: Fluzone® (Aventis Pasteur inactivated influenza vaccine)
- Male, Age 50 -64, Half Dose (Experimental): 0.25ml, 7.5µg Fluzone® (Aventis Pasteur inactivated influenza vaccine) hemagglutinia per strain
  Interventions: Biological: Fluzone® (Aventis Pasteur inactivated influenza vaccine)
- Female, Age 18 - 49, Full Dose (Experimental): 0.5ml, 15µg Fluzone® (Aventis Pasteur inactivated influenza vaccine) hemagglutinin antigen per strain
  Interventions: Biological: Fluzone® (Aventis Pasteur inactivated influenza vaccine)
- Female, Age 18 - 49, Half Dose (Experimental): 0.25ml, 7.5µg Fluzone® (Aventis Pasteur inactivated influenza vaccine) hemagglutinia per strain
  Interventions: Biological: Fluzone® (Aventis Pasteur inactivated influenza vaccine)
- Male, Age 18 - 49, Half Dose (Experimental): 0.25ml, 7.5µg Fluzone® (Aventis Pasteur inactivated influenza vaccine) hemagglutinia per strain
  Interventions: Biological: Fluzone® (Aventis Pasteur inactivated influenza vaccine)
- Male, Age 50 -64, Full Dose (Experimental): 0.5ml, 15µg Fluzone® (Aventis Pasteur inactivated influenza vaccine) hemagglutinin antigen per strain
  Interventions: Biological: Fluzone® (Aventis Pasteur inactivated influenza vaccine)
- Female, Age 50 -64, Full Dose (Experimental): 0.5ml, 15µg Fluzone® (Aventis Pasteur inactivated influenza vaccine) hemagglutinin antigen per strain
  Interventions: Biological: Fluzone® (Aventis Pasteur inactivated influenza vaccine)
- Female, Age 50 -64, Half Dose (Experimental): 0.25ml, 7.5µg Fluzone® (Aventis Pasteur inactivated influenza vaccine) hemagglutinin antigen per strain
  Interventions: Biological: Fluzone® (Aventis Pasteur inactivated influenza vaccine)

INTERVENTIONS:
Biological: Fluzone® (Aventis Pasteur inactivated influenza vaccine) — A/H1N1, A/New Caledonia/20/99; A/H3N2, A/Fujian/411/2002; B, B/Shanghai/361/2002

SUMMARY:
This study compared full-dose Flu vaccine to half-dose Flu-vaccine during the 2004-2005 flu season.

DETAILED DESCRIPTION:
This was a Phase II prospective, single-blind to dose, randomized study that compared the immunogenicity of subjects receiving half-dose Fluzone® compared to full-dose Fluzone®, 2004-2005 formulation. 1440 healthy subjects, ages 18-64 years old and not currently indicated for influenza vaccination under the interim ACIP guidelines, were divided into 8 strata based on age, gender, and previous exposure to influenza vaccine, and randomized to receive either half-dose (0.25mL) Fluzone® or full-dose (0.5mL) Fluzone® by intramuscular injection into the deltoid muscle.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and comply with all study procedures including availability for all study visits and follow up surveys within 6 months following study enrollment.
* DEERS eligible beneficiaries eligible for influenza vaccination and able to give informed consent.
* Age 18-49

  * Patients presenting to travel clinic with no exclusion criteria;
  * Household contacts and out-of-home caretakers of infants from 6-23 months of age;
  * Hospital and/or employees providing service to the public who are not eligible for the post-October 5th recommendations for priority immunization;
  * DOD employees eligible for influenza vaccination prior to October 5th but excluded in the post October 5th guidelines;
  * People living in dormitories or under other crowded conditions, to prevent outbreaks;
* Ages 50-64 years of age who are not eligible for the post-October 5th recommendations for priority immunization and with no standard of care contraindications to vaccination.
* Eligible in the Department of Defense for influenza vaccination

Exclusion Criteria:

* all children aged < 18 years (includes children aged 6 months-18 years on chronic aspirin therapy);
* adults aged >65 years;
* persons aged 2-64 years with underlying chronic medical conditions:

  * includes persons with chronic cardiac or pulmonary disease, diabetes mellitus, hemoglobinopathy, or immunosuppressive illness;
  * any acute or chronic condition that, in the opinion of the investigator, would render vaccination unsafe or interfere with the evaluation of response.
* use of experimental vaccines or medications within 30 days of study entry;
* receipt of parenteral immunoglobulin within 60 days of study entry;
* all women who will be pregnant during the influenza season;
* residents of nursing homes and long-term care facilities;
* health-care workers involved in direct patient care and included in DOD priority 1; and;
* military recruits;
* out-of-home caregivers and household contacts of children aged <6 months.
* Anyone with clinical contraindications for receiving the inactivated influenza vaccine such as a history of severe allergic reaction to prior influenza vaccinations, severe allergy to egg and/or egg proteins and gelatin.
* DOD Priority 1: Deployed or deploying (with orders) service members and others designated as critical to national defense.
* DOD Priority 2: Medically high risk in accordance with ACIP guidelines (includes health-care workers with direct patient contact)
* Any acute or chronic condition that, in the opinion of the investigator or her provider designee would render vaccination unsafe or interfere with the evaluation of the response.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1316 (Actual)
Dates: Start 2004-11 (Actual); Primary Completion 2004-11 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renata J Engler, M.D, Principal Investigator — Walter Reed Army Medical Center
Locations (2):
- United States (2):
  - Pentagon, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Engler RJ, Nelson MR, Klote MM, VanRaden MJ, Huang CY, Cox NJ, Klimov A, Keitel WA, Nichol KL, Carr WW, Treanor JJ; Walter Reed Health Care System Influenza Vaccine Consortium. Half- vs full-dose trivalent inactivated influenza vaccine (2004-2005): age, dose, and sex effects on immune responses. Arch Intern Med. 2008 Dec 8;168(22):2405-14. doi: 10.1001/archinternmed.2008.513. PMID 19064822

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited at the Walter Reed Army Medical Center Allergy-Immunization Clinic, the Fort Belvoir DeWitt Allergy-Immunization Clinic and the Pentagon Health Clinic during the annual influenza immunization program.
Pre-assignment Details: Enrollment was expanded to include subs with a history of flu vacs. From the originally enrolled subjects (1316), the final data analysis includes only members of the baseline re-vaccination population (1114).
Groups:
- Full Dose, Age 18-49: Subjects age 18-49 receiving full dose
- Half Dose, Age 18-49: Subjects age 18-49 receiving half dose
- Full Dose, Age 50-64: Subjects age 50-64 receiving full dose
- Half Dose, Age 50-64: Subjects age 50-64 receiving half dose
Period: Overall Study
Arm/Group | Full Dose, Age 18-49 | Half Dose, Age 18-49 | Full Dose, Age 50-64 | Half Dose, Age 50-64
Started | 274 | 284 | 280 | 276
Completed | 274 | 284 | 280 | 276
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: FCSR didn't report baseline demographics per arm they were presented by age group.
Groups:
- Full Dose, Age 18-49: Previously Vaccinated Subjects Receiving Full Dose Aged 18-49 Years
- Half Dose, Age 18-49: Previously Vaccinated Subjects Receiving Half Dose Aged 18-49 Years
- Full Dose, Age 50-64: Previously Vaccinated Subjects Receiving Full Dose Aged 50-64 Years
- Half Dose, Age 50-64: Previously Vaccinated Subjects Receiving Half Dose Aged 50-64 Years
- Total: Total of all reporting groups
Arm/Group | Full Dose, Age 18-49 | Half Dose, Age 18-49 | Full Dose, Age 50-64 | Half Dose, Age 50-64 | Total
Number analyzed (Participants) | 274 | 284 | 280 | 276 | 1114
Age, Customized [Number; unit: years] | 274 | 284 | 280 | 276 | 1114
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 121 | 119 | 118 | 484
  Male | 148 | 163 | 161 | 158 | 630
Region of Enrollment [Number; unit: participants]
  United States | 274 | 284 | 280 | 276 | 1114

OUTCOME MEASURES:

1. Primary Outcome: Immune Response: Age 18-49
Description: Immune response as measured by viral strain specific hemaggluttination inhibition (HAI) antibody levels for subjects ages 18-49
Time Frame: 21 days post-vaccincation
Population: From the 1263 subjects enrolled, final analysis includes baseline re-vaccinated subs who fit all inc/exc criteria and whose serum specimens were usable. Data summarizes the differences in influenza strain specific serologic responses according to vaccine dose and age. Antibodies were measured by Hemagglutination Inhibition. GMT=Geometric Mean Titer
Measure: Geometric Mean (95% Confidence Interval); unit: Anti-body response (GMT)
Groups:
- Age 18 - 49, Full Dose: 0.5ml, 15µg Fluzone® (Aventis Pasteur inactivated influenza vaccine) hemagglutinin antigen per strain
  Fluzone® (Aventis Pasteur inactivated influenza vaccine): A/H1N1, A/New Caledonia/20/99; A/H3N2, A/Fujian/411/2002; B, B/Shanghai/361/2002
- Age 18 - 49, Half Dose: 0.25ml, 7.5µg Fluzone® (Aventis Pasteur inactivated influenza vaccine) hemagglutinia per strain
  Fluzone® (Aventis Pasteur inactivated influenza vaccine): A/H1N1, A/New Caledonia/20/99; A/H3N2, A/Fujian/411/2002; B, B/Shanghai/361/2002
Arm/Group | Age 18 - 49, Full Dose | Age 18 - 49, Half Dose
Number analyzed (Participants) | 274 | 284
Anti-body response (GMT)
  H1N1 - GMT | 28.8 [25.2 to 32.8] | 21.3 [18.9 to 24.0]
  H3N2 - GMT | 55.2 [48.7 to 62.5] | 45.0 [39.7 to 50.9]
  B - GMT | 69.6 [61.4 to 78.9] | 54.8 [49.1 to 61.2]

2. Primary Outcome: Immune Response: Age 50-64
Description: Immune response as measured by viral strain specific hemaggluttination inhibition (HAI) antibody levels for subjects ages 50-64
Time Frame: 21 days post-vaccincation
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Anti-body response (GMT)
Groups:
- Age 50 - 64, Full Dose: 0.5ml, 15µg Fluzone® (Aventis Pasteur inactivated influenza vaccine) hemagglutinin antigen per strain
  Fluzone® (Aventis Pasteur inactivated influenza vaccine): A/H1N1, A/New Caledonia/20/99; A/H3N2, A/Fujian/411/2002; B, B/Shanghai/361/2002
- Age 50 - 64, Half Dose: 0.25ml, 7.5µg Fluzone® (Aventis Pasteur inactivated influenza vaccine) hemagglutinia per strain
  Fluzone® (Aventis Pasteur inactivated influenza vaccine): A/H1N1, A/New Caledonia/20/99; A/H3N2, A/Fujian/411/2002; B, B/Shanghai/361/2002
Arm/Group | Age 50 - 64, Full Dose | Age 50 - 64, Half Dose
Number analyzed (Participants) | 280 | 276
Anti-body response (GMT)
  H1N1 - GMT | 21.4 [18.6 to 24.7] | 14.2 [12.7 to 15.9]
  H3N2 - GMT | 59.0 [51.4 to 67.8] | 39.1 [34.3 to 44.6]
  B - GMT | 52.1 [45.5 to 59.8] | 36.8 [32.4 to 41.9]

3. Secondary Outcome: Medical Events: Unsolicited Adverse Events
Description: Assessed through following subjects' recording of oral body temperature, completion of a 21-day symptom diary; subjects' completion of longer-term follow-up surveys to track respiratory symptoms; and a review of the Defense Medical Surveillance System (DMSS) hospitalization and outpatient medical visits database in order to track ICD-9 codes relevant to flu-like illness.
Time Frame: 3 - 6 months following vaccination
Population: Of the original population, 1203 previously vaccinated subjects completed the 3-day post vaccination side effects diary and have been included in the this analysis.
Measure: Number; unit: Adverse events
Groups:
- Mild: Mild AE
- Moderate: Moderate AE
- Severe, Able to Work: Severe but able to work
- Severe, Lost Productivity: Severe and lost productivity
- No Events: No adverse events recorded
Arm/Group | Mild | Moderate | Severe, Able to Work | Severe, Lost Productivity | No Events
Number analyzed (Participants) | 1203 | 1203 | 1203 | 1203 | 1203
Adverse events
  Body as a Whole | 0 | 6 | 1 | 3 | 1193
  Cardiovascular System | 2 | 2 | 0 | 0 | 1199
  Digestive Sytem | 12 | 3 | 2 | 4 | 1182
  Hematological and Lymphatic System | 2 | 0 | 1 | 0 | 1200
  Musculoskeletal System | 6 | 5 | 1 | 1 | 1190
  Respiratory System | 10 | 18 | 5 | 3 | 1167
  Skin and Appendages | 14 | 8 | 1 | 0 | 1180
  Special Senses | 2 | 2 | 0 | 1 | 1198
  Urogenital System | 0 | 4 | 0 | 0 | 1199
  Symptions in Arm Given Shot | 13 | 1 | 0 | 0 | 1189
  Headache | 0 | 2 | 1 | 1 | 1199

4. Other Pre Specified Outcome: Race/Ethnicity Baseline Measure
Description: Race/ethnicity data was only collected by age and cannot be separated out by dose as per the other Baseline Measures
Time Frame: Enrollment Day
Measure: Count of Participants; unit: Participants
Groups:
- Aged 18-49 y (n=558): Race/Ethnicity stratified by age 18-49
- Aged 50-64 y (n=556): Race/Ethnicity stratified by age 50-64
Arm/Group | Aged 18-49 y (n=558) | Aged 50-64 y (n=556)
Number analyzed (Participants) | 558 | 556
Participants
  White | 454 | 491
  African American | 54 | 46
  Hispanic | 16 | 6
  Asian | 14 | 7
  Other/unknown | 10 | 6

ADVERSE EVENTS:
Time Frame: 3 - 6 months following vaccination
Description: Of the original study population, 1203 previously vaccinated subjects completed the 3-day post vaccination side effects diary and have been included in this analysis.
  AEs were collected with diary cards, health surveys, and VAERS forms and listed by subject
  Grading of AE's:
  1 = Mild; 2 = Moderate; 3 = Severe, able to work; 4 = Severe, lost productivity; 5 = Life-threatening; 6 = Fatal
Groups:
- Full Dose: 0.5ml, 15µg Fluzone® (Aventis Pasteur inactivated influenza vaccine) hemagglutinin antigen per strain
  Fluzone® (Aventis Pasteur inactivated influenza vaccine): A/H1N1, A/New Caledonia/20/99; A/H3N2, A/Fujian/411/2002; B, B/Shanghai/361/2002
- Half Dose: 0.25ml, 7.5µg Fluzone® (Aventis Pasteur inactivated influenza vaccine) hemagglutinia per strain
  Fluzone® (Aventis Pasteur inactivated influenza vaccine): A/H1N1, A/New Caledonia/20/99; A/H3N2, A/Fujian/411/2002; B, B/Shanghai/361/2002
Arm/Group | Full Dose | Half Dose
All-Cause Mortality (participants affected / at risk) | 0/554 | 0/556
Serious Adverse Events (participants affected / at risk) | 2/554 | 1/556
Other Adverse Events (participants affected / at risk) | 18/554 | 17/556
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Dose (N=554) | Half Dose (N=556)
Carotid endarterectomey (Cardiac disorders) | 0 (0) | 1 (1)
Melanoma exised (Surgical and medical procedures) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Dose (N=554) | Half Dose (N=556)
Brusing at injection site (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) — Grade 1
Body aches (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Grade 2
Bruising at injection site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Grade 3
Aching at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Grade 1
Arm sore at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Grade 1
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) — Grade 1
Fever, chills, flu-like symptoms (General disorders) | 1 (1) | 0 (0) — Grade 4
Flu-like symptoms (General disorders) | 0 (0) | 1 (1) — Grade 4
Flu-like symptoms (General disorders) | 0 (0) | 1 (1) — Grade 2
Hurt at injection site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Grade 2
Idiopathic urticaria (Immune system disorders) | 0 (0) | 1 (1) — Grade 1
Ichiness at injection site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Grade 1
Injection site soreness (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) — Grade 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) — Grade 4
Itching, distil to injection site (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — Grade 1
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 1
Nausea and body aches (Gastrointestinal disorders) | 0 (0) | 1 (1) — Grade 4
Outbreak of HSV on face, also nasal lesions (Infections and infestations) | 1 (1) | 0 (0) — Grade 2
Pain in right antecubital area after venipuncture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Grade 1
Rash on right calf (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Grade 2
Right shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Grade 1
Sore, achy shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Grade 2
Swollen lymph nodes (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Grade 1
Swollen lymph nodes in neck, sore throat, chills, body aches (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Grade 1
Tender at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Grade 1
Tingling in fingers of vaccinated arm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Grade 1
Very sore at injection site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Grade 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No